CLINICAL TRIAL: NCT07254234
Title: Exploratory Study to Assess Utility of RetiSpec Artificial Intelligence Powered Retinal Imaging Solution in Detecting Amyloid Pathology in United Arab Emirates Nationals With Mild Impairment of Cognition
Brief Title: A Study of Retinal Imaging to Detect Abnormal Protein Deposits Associated With Alzheimer's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 27414; H7I-MC-S035 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Dysfunction; Memory Disorders
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Memory Complaints or Mild Cognitive Impairment (MCI): Retinal scan and blood biomarker testing
  Interventions: Other: Retinal scan; Other: Blood test

INTERVENTIONS:
Other: Retinal scan — Detailed image of the retina.
Other: Blood test — Sample will be used to test for a specific form of a protein in the blood to learn more about early detection of Alzheimer's disease.

SUMMARY:
The purpose of this study is to test the use of a screening tool to detect changes in the eye that are associated with Alzheimer's disease in adult participants with memory issues. For each participant, the study will last up to one month and requires one visit to the research site.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including medical history and physical examination.
* Have mild memory complaints or a diagnosis of mild cognitive impairment.
* Have undergone genotyping for apolipoprotein E (APOE) and are willing to make results available to the investigator.
* Montreal Cognitive Assessment (MoCA) score of greater than or equal to 22 and less than or equal to 28.

Exclusion Criteria:

* Have any medical condition that, in the opinion of the investigator, would be a contraindication to participation in the study.
* Have an existing diagnosis of AD or other dementia.
* Have contradictions to or an allergy to the ophthalmic dilating agents.
* Have known diagnosis of severe glaucoma or severe cataracts; have a significant refractive error (more than 12 diopters [D] of spherical equivalent refraction); or have any ocular media opacity that prevents imaging of the retina (that is, severe cataract). Note: mild to moderate cataracts or vision correction with glasses or contact lenses are not exclusion criteria.
* Current or previous treatment with anti-amyloid medications.
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emiratis age 55 or older with mild memory complaints or MCI who are otherwise healthy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with the Same Results on the Blood Test and Retinal Scan | Day 1

SECONDARY OUTCOMES:
Percentage of Participants who Report High or Moderate Satisfaction with Retinal Scan | Day 1
  Measured by 5-item retinal scan feedback survey. Participants rate their experience with the retinal scan on a 5-item Likert scale that ranges from "Strongly Disagree" to "Strongly Agree." Higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No